CLINICAL TRIAL: NCT02451488
Title: Neoadjuvant GM-CSF Treatment and Modulation of Immune Cell Profile of the SLN in Melanoma
Brief Title: Neoadjuvant Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Cutaneous Stage L-lll Melanoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James W. Jakub, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-005510
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GM-CSF (Experimental): Patients will be treated with 14 days of GM-CSF self-administered subcutaneously daily for 14 days in a dose of 125 µg/m2 beginning on the day of enrollment. Patients will be instructed in the self-administration of GM-CSF and after they have demonstrated competency with the procedure, they will self-administer the treatment at home. Patients will undergo surgery within 1 day to 5 days after cessation of the GM-CSF therapy.
  Interventions: Drug: GM-CSF
- Standard of Care (Other): no neo-adjuvant therapy prior to surgical intervention
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: GM-CSF — 14 days in a dose of 125 µg/m^2
  Other Names: Leukine
  Arms: GM-CSF
Other: Standard of Care — No neo-adjuvant therapy prior to surgical intervention
  Arms: Standard of Care

SUMMARY:
Randomized trial to determine if neo-adjuvant subcutaneous GM-CSF restores the host regional lymph node immunity

DETAILED DESCRIPTION:
The sentinel lymph nodes in patients with melanoma are immunosuppressed and the investigators have shown this occurs early in the disease process. This regional nodal immunosuppression precedes nodal metastasis and may be required for nodal spread. Administration of GM-CSF has been used to alter the immune response to metastatic melanoma. The investigators propose to assess whether administration of a short course of GM-CSF preoperatively to patients about to undergo wide local excisions and sentinel lymph node dissection can alter the immune environment of the sentinel lymph node and restore an immune surveillance profile in the sentinel lymph node.

ELIGIBILITY:
Inclusion Criteria

To be eligible for the study, patients must satisfy the following criteria:

* Histologically confirmed primary cutaneous malignant melanoma
* 1-4mm Breslow depth
* Scheduled for sentinel lymph node biopsy as part of their standard surgical management
* Man or woman, age >/= 18 years
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 2 weeks after the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal. Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. All WOCBP must have a negative pregnancy test prior to first receiving GM-CSF.
* Men must agree to use and utilize an adequate method of contraception throughout treatment and for at least 2 weeks after study drug is stopped
* All patients must be willing and able to give written informed consent.

Exclusion Criteria Subjects meeting any of the following criteria are ineligible for study entry

* Clinical stage III or IV disease
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of immunologic disease (e.g. rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis, motor neuropathy considered of autoimmune origin)
* Any underlying medical conditions which, in the opinion of the investigator, will make the administration of GM-CSF hazardous or obscure the interpretation of adverse events; such as, psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and followup schedule
* Any vaccination therapy within 4 weeks prior to GM-CSF administration
* Concomitant therapy with any of the following within the past 3 months: GM-CSF, interferon, other non-study immunotherapy regimes; cytotoxic chemotherapy
* Immunosuppressive mediations (steroids, tumor necrosis factor (TNF)-inhibitors, azathioprine, etc.) within the past 6 weeks
* Active or chronic infection with HIV, hepatitis B or hepatitis C
* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and 2 weeks after cessation of the study drug.
* Prisoners or subjects who are compulsorily detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Jakub, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
data will not be shared

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GM-CSF | Standard of Care
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GM-CSF | Standard of Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.3) | 62.7 (18.8) | 58.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Th1/Th2 Normalized Gene Expression
Description: The Th1/Th2/Th3 Reverse transcription polymerase chain reaction (RT-qPCR) arrays will be used to quantify RNA expression of Th1 and Th2 messenger ribonucleic acids (mRNAs). Normalized gene expression was calculated from qRT-PCR results comparing GM-CSF and control subjects for both Th1-associated gene T-bet and Th2-associated gene GATA3 respectively. Fold change values are calculated by taking the normalized gene expression in GM-CSF treated group samples divided by the normalized gene expression in the control group samples.
Time Frame: 14 days post treatment
Population: Three subjects were in in the GM-CSF group and three subjects were in the Standard of Care group. One subject in the GM-CSF group received GM-CSF but did not have tissue sample collected for research analysis. One subject in the Standard of Care group did not have a large enough tissue sample collected to be analyzed.
Measure: Mean (95% Confidence Interval); unit: fold change
Groups:
- Standard of Care: no neo-adjuvant therapy prior to surgical intervention Standard of Care: No neo-adjuvant therapy prior to surgical intervention
Arm/Group | GM-CSF | Standard of Care
Number analyzed (Participants) | 3 | 3
fold change
  T-bet (Th1) | 1.029 [0.999 to 1.059] | 0.119 [-1.506 to 1.654]
  GATA3 (Th2) | 0.074 [-0.041 to 0.279] | 0.192 [0.068 to 0.316]

ADVERSE EVENTS:
Time Frame: 14 days
Description: Subjects receiving intervention will have adverse events (AEs) recorded during the 14 day course of self-administrated GM-CSF. Subjects will be provided a diary to record any AEs. Subjects will be provided a list of AEs and to call immediately for any grade 3 or high AEs. Grade I-II AEs will be logged into their diary. Diary will be collected the day of surgery. All-Cause Mortality, Serious, and Other (Not Including Serious) AEs were not monitored/assessed for the Standard of Care Arm/Group.
Arm/Group | GM-CSF | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02451488/Prot_SAP_000.pdf